CLINICAL TRIAL: NCT02513108
Title: Stavanger UncomPlicatEd Elective PCI Same DaY Discharge Study (SPEEDY Study)
Acronym: SPEEDY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SUS2015NIBO01
Record Dates: First submitted 2015-07-17; First posted 2015-07-31 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Masking Description: original sample size calculation is amended from 151 patients to 82 patients after recalculation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- same day discharge (Active Comparator): patients discharged same day after uncomplicated PCI
  Interventions: Procedure: same day discharge
- standard care (No Intervention): standard care where patients are discharged the day after procedure after adequate observation

INTERVENTIONS:
Procedure: same day discharge — same day discharge after PCI for stable CAD
  Arms: same day discharge

SUMMARY:
The purpose of this study is to provide information on safety of same day discharge after uncomplicated percutaneous intervention (PCI) for stable angina pectoris in Norwegian clinical practice. The investigators also think that is in patients interest to stay as short time as possible in hospital and this will be measured using standardised quality of life questionnaires.

DETAILED DESCRIPTION:
The international literature has already provided documentation on the safety of same day discharge in various clinical scenario. In this particular study, the investigators focus on challenging the contemporary Norwegian practice where every body stays over night.

Only patients with stable angina pectoris will be included in the study. After informed consent and successful procedure, the patients will be randomised to same day discharge or standard care. Same day discharge patients will be contacted by telephone the day after the procedure for follow-up conversation with particular emphasis on access site complications.

Both groups will receive quality of life questionnaire within a month for assessment of difference between the two strategies.

ELIGIBILITY:
Inclusion Criteria:

* Elective procedures Monday through Thursday
* Patient consenting for same day discharge
* Operator has assessed the patient and is in agreement
* Adequate observational facility
* Uncomplicated procedure
* Acceptable social network at home
* Uneventful post PCI ECG
* Adequate hemostasis of puncture site

Exclusion Criteria:

* Angiographic

  * No-reflow/slow flow post PCI
  * Sub-optimal PCI result
  * Dissection type C-E
  * Rest dissection after stent deployment
  * Angiographic thrombus
  * Guidewire perforation
* Clinical

  * Advanced age
  * Severe renal failure (GFR < 30ml/min)
  * Excessive bleeding risk
  * Symptomatic heart failure
  * Severe visual or hearing impairment
  * Multi-vessel PCI (2 main vessels or left main)
  * Use of GP IIb/IIIa inhibitors
* Social

  * Living alone or has no telephone
  * Long driving distance (> 30-45 min)
  * Patient/next to keen can´t communicate with health personnel without a translator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
number of complications (access site bleeding) | 1 month
  observation of complications requiring intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nigussie Bogale, M.D, PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: No